CLINICAL TRIAL: NCT06291441
Title: Female Urinary Incontinence in Middle-aged Women in Four Hospitals in Northern Italy: a Multicenter Prevalence Study
Brief Title: Women Urinary Incontinence Prevalence Study (WUIPS)
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Sara Trapani, Principal Investigator, Midwife (RM), PhD student, IRCCS San Raffaele
Other Study IDs: WUIPS
Record Dates: First submitted 2024-02-16; First posted 2024-03-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Female Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women's single sample: INSTRUMENTS:
  * UI Survey: A survey, written in Italian by the authors, will collect women's socio-demographic, economic and clinical characteristics
  * Italian version of International Consultation of Incontinence Modular Questionnaire Urinary Incontinence Short Form (ICIQ UI-SF)
  * Italian version of Incontinence Impact Questionnaire-7 (IIQ-7)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention (observational study)

SUMMARY:
The goal of this multicenter prospective and prevalence observational study is to punctually investigate and describe prevalence, predictors, quality of life and costs of Urinary Incontinence (UI) among female patients, female caregivers and female personnel in four hospitals in Northern Italy: San Raffaele hospital in Milan, San Raffaele Turro hospital in Milan, Zingonia Policlinico San Marco (BG) and Policlinico San Pietro in Ponte San Pietro (BG).

DETAILED DESCRIPTION:
EXPECTED RESULTS

The collection of data and information through this study will aim to:

1. Understand the percentage of middle-aged women with UI.
2. Describe the socio-demographic and clinical characteristics of women with UI.
3. Identify UI predictors.
4. Describe the quality of life, social impact and costs of women with UI.

ELIGIBILITY:
INCLUSION CRITERIA

* Female sex
* Middle age (40-65 years old)
* Informed consent signed
* Comprehension of written and spoken Italian language
* Female outpatients intended for any hospital unit (outpatient clinic, day surgery and day hospital patients included) and every female caregiver respecting the previous inclusion criteria, recruited at the central admission and at the private admission of the four hospitals involved
* Female workers (healthcare professionals and administrative personnel) of the four hospitals

EXCLUSION CRITERIA

* Male sex
* Young age (< 40 years) and older age (> 65 years)
* Pregnant women
* Puerperium women (up to 40 days post-partum)
* Women who had undergone urinary and gynecology surgery

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All female patients, female caregivers, female healthcare professionals and female administrative workers who meet the inclusion criteria will be included. Participants will be enrolled in four centers in Northern Italy which are the reference centers for UniSR: San Raffaele hospital in Milan, San Raffaele Turro hospital in Milan, Zingonia Policlinico San Marco (BG) and Policlinico San Pietro in Ponte San Pietro (BG).
Sampling Method: Non-Probability Sample
Enrollment: 449 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of middle-aged women with urinary incontinence | by December 2025
  Epidemiological data
  Measure:
  - Italian version of International Consultation of Incontinence Modular Questionnaire Urinary Incontinence Short Form (ICIQ UI-SF)

SECONDARY OUTCOMES:
Predictors of urinary incontinence in middle-aged women | by December 2025
  Description and association between UI and related predictors
  Measure:
  - UI Survey: A part of the survey, written in Italian by the authors, will collect women's socio-demographic and clinical characteristics (predictors of UI)
Quality of life of middle-aged women with urinary incontinence | by December 2025
  Description and association between UI and quality of life
  Measure:
  - Italian version of Incontinence Impact Questionnaire-7 (IIQ-7) for investigating women's quality of life
Social impact of middle-aged women with urinary incontinence | by December 2025
  Description and association between UI and social impact
  Measure:
  - UI Survey: A part of the survey, written in Italian by the authors, will collect social impact of UI through a 4-point Likert scale
Costs of urinary incontinence for middle-aged women | by December 2025
  Description of UI costs
  Measure:
  - UI Survey: A part of the survey, written in Italian by the authors, will collect costs of UI through a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Duilio F. Manara, Study Director — Director of Center for Nursing Research and Innovation (CeNRI); Stefano Salvatore, Study Director — U.O. Obstetrics and Gynecology; Massimo Candiani, Study Director — Director of U.O. Obstetrics and Gynecology
Locations (4):
- Italy (4):
  - Policlinico San Marco Zingonia, Osio Sotto, Bergamo
  - Policlinico San Pietro Ponte San Pietro, Bergamo
  - San Raffaele Turro Hospital (MI), Milan
  - San Raffaele Hospital (MI), Milan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT06291441/Prot_000.pdf